CLINICAL TRIAL: NCT04546620
Title: A Randomised Phase II Evaluation of Molecular Guided Therapy for Diffuse Large B-Cell Lymphoma With Acalabrutinib
Brief Title: Acalabrutinib in Combination With R-CHOP for Previously Untreated Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: REMoDL-A
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM CAN1500
Record Dates: First submitted 2020-08-11; First posted 2020-09-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Lymphoma; Acalabrutinib; R-CHOP; DLBCL; Non Hodgkin Lymphoma; Haematological cancer; Bruton Tyrosine Kinase; Molecular Profiling; Chemoimmunotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin | interventions — R-CHOP protocol; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A Control (Active Comparator): 6 cycles of standard R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisolone) immunochemotherapy every 21 days.
  Interventions: Drug: R-CHOP
- Arm B Experimental (Experimental): 1 cycle of standard R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisolone) immunochemotherapy followed by 5 cycles of R-CHOP + acalabrutinib taken twice daily for 21 day cycles.
  Interventions: Drug: R-CHOP + acalabrutinib

INTERVENTIONS:
Drug: R-CHOP — Arm A patients will receive R-CHOP alone.
  Other Names: Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone
  Arms: Arm A Control
Drug: R-CHOP + acalabrutinib — Arm B patients will receive R-CHOP in combination with acalabrutinib.
  Other Names: Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Acalabrutinib
  Arms: Arm B Experimental

SUMMARY:
This study evaluates the addition of Acalabrutinib to current standard therapy of Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisolone (R-CHOP) for patients with previously untreated CD20 positive Diffuse Large B-cell Lymphoma (DLBCL) requiring full course chemoimmunotherapy.

All patients will receive one cycle of R-CHOP. Two thirds of patients (Arm B) will go on to receive a further 5 cycles (every 21 days) of R-CHOP with Acalabrutinib. Acalabrutinib will be taken orally twice daily continuously in 21 day cycles.

One third of patients (Arm A) will continue with 5 cycles of R-CHOP.

Patients will be followed up initially for 24 months and then for disease status and survival until 114 progression events have been observed.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common of the non-Hodgkin's lymphomas. Whilst the majority of patients will respond well to conventional treatment (R-CHOP - rituximab, cyclophosphamide, doxorubicin, vincristine and prednisolone), a significant number of patients lymphoma will not respond to initial therapy or their disease will return after completion of therapy. In a number of B-cell diseases an enzyme called, Bruton tyrosine kinase (BTK) prevents death of tumour cells, including in DLBCL. Acalabrutinib is an orally active BTK-inhibitor and it is thought that stopping BTK being activated may help in treating B-cell diseases. It is hypothesised that the addition of Acalabrutinib to standard R-CHOP immunochemotherapy may improve outcomes of patients with DLBCL.

REMoDL-A is a randomised, phase II, open label, multicentre study that will be open in up to 50 centres. Up to 553 patients (453 randomised) will be recruited.

Following informed consent all patients will receive 1 cycle of conventional R-CHOP chemotherapy. At the same time the diagnostic pathology block will be sent for molecular profiling by the Haematological Malignancy Diagnostic Service (HMDS). The delivery of the first cycle of R-CHOP will allow a sufficient interval for real time determination of molecular phenotype. Patients whose biopsies yield sufficient tumour material for profiling will be randomised 2:1 in favour of the experimental arm (R-CHOP + acalabrutinib).

The primary objective will be to establish if combining acalabrutinib with R-CHOP improves efficacy, compared to R-CHOP alone, for the treatment of previously untreated patients with DLBCL to a degree that justifies further development of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL, expressing CD20. Sufficient diagnostic material must be available to forward to HMDS for gene expression profiling and central pathology review. The following diagnoses by 2016 WHO classification of lymphoid neoplasms may be included:

  * DLBCL, not otherwise specified (NOS)
  * T-cell/histiocyte-rich large B-cell lymphoma
  * Epstein-Barr virus positive DLBCL, NOS
  * ALK-positive large B-cell lymphoma
  * HHV8-positive DLBCL, NOS
  * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (double-hit or triple-hit lymphoma)
  * High-grade B-cell lymphoma, NOS
* At least one bi-dimensionally measurable lesion, defined as >1.5 cm in its longest dimension as measured by CT.
* Not previously treated for lymphoma and fit enough to receive combination chemoimmunotherapy with curative intent.
* Stage IAX (bulk defined as lymph node mass [either single or conglomerate] diameter >7.5cm) to stage IV disease and deemed to require a full course of chemotherapy. Patients with non-bulky IE disease will not be eligible.
* ECOG performance status 0-2 or 3 if this is directly attributable to lymphoma.
* Adequate bone marrow function with platelets > 100x109/L; neutrophils > 1.0x109/L at study entry, unless lower figures are attributable to lymphoma.
* Measured or calculated creatinine clearance > 30mls/min, (calculated using the formula of Cockcroft and Gault [(140-Age) x Mass (kg) x (1.04 (for women) or 1.23 (for men))/Serum Creatinine (μmolL)]).
* Serum bilirubin < 35μmol/L and transaminases < 1.5x upper limit of normal at time of study entry.
* Cardiac function sufficient to tolerate 300mg/m2 of doxorubicin. A pre-treatment echocardiogram or MUGA is required to establish baseline LVEF equal to or greater than institutional normal range.
* No concurrent uncontrolled medical condition.
* Life expectancy > 3 months.
* Aged 16 years or above.
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent.

Exclusion Criteria:

* Previous history of treated or untreated indolent lymphoma. However newly diagnosed patients with DLBCL who are found to also have small cell infiltration of the bone marrow or other diagnostic material (discordant lymphoma) will be eligible.
* Patients who have received immunisation with a live vaccine within four weeks prior to enrolment will be ineligible.
* Diagnosis of primary mediastinal lymphoma.
* Diagnosis of primary Central Nervous System lymphoma or secondary CNS involvement. Those patients presenting with neurological symptoms should be investigated for CNS involvement. Routine CNS imaging or diagnostic lumbar puncture will not be required in the absence of symptoms.
* History of stroke or intracranial haemorrhage in preceding 6 months.
* History of bleeding diathesis (eg, haemophilia, von Willebrand disease).
* History of drug-specific hypersensitivity or anaphylaxis to any study drug (including active product or excipient components).
* Requires or receiving anticoagulation with warfarin or equivalent antagonists (eg, phenprocoumon) within 7 days of first dose of acalabrutinib. However patients using therapeutic low molecule weight heparin or low dose aspirin will be eligible as will those receiving direct oral anticoagulants.
* Prior exposure to an inhibitor in the BCR pathway (eg, Btk inhibitors, phosphoinositide-3 kinase (PI3K), or Syk inhibitors) or BCL-2 inhibitor (eg, ABT-199).
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
* Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Patients receiving proton pump inhibitors should switch to short-acting H2-receptor antagonists or antacids prior to the commencement of acalabrutinib, if randomised to receive acalabrutinib.
* Active significant infection (e.g. progressive multifocal leukoencephalopathy (PML)).
* Uncontrolled autoimmune haemolytic anaemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
* Major surgery in the preceding 4 weeks of first dose of acalabrutinib (if applicable). If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of acalabrutinib (if applicable).
* Corticosteroid use >30 mg/day of prednisone or equivalent, for purposes other than for lymphoma symptom control. Patients receiving corticosteroid treatment with <30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to the start of Cycle 1. If glucocorticoid treatment is urgently required for lymphoma symptom control prior to the start of study treatment, prednisone 100 mg or equivalent could be given for a maximum of 14 days as a prephase. A dose of up to 30mg or prednisolone or equivalent may be used during the screening phase to control symptoms.
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
* Serological positivity for Hepatitis B, C, or known HIV infection. As per standard of care, prior to initiation of immunochemotherapy, the results of hepatitis serology should be known prior to commencement of therapy.

  1. Positive test results for chronic HBV infection (defined as positive HBsAg serology) will not be eligible. Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) will not be eligible. Patients who have protective titres of hepatitis B surface antibody (HBsAb) after vaccination will be eligible.
  2. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Women who can bear children must agree to use two highly effective forms of contraception or abstinence during the study and for 12 months after the last treatment dose.
* Breastfeeding or pregnant women.
* Men who can father children must agree to use two highly effective forms of contraception with additional barrier or abstinence during the study and for 12 months after the last treatment dose.
* Men must agree to refrain from sperm donation during the study and for 12 months after the last treatment dose.
* Serious medical or psychiatric illness likely to affect participation or that may compromise the ability to give informed consent.
* Prior malignancy (other than DLBCL), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years.
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease, resection of the stomach or small bowel, partial or complete bowel obstruction or gastric restrictions and bariatric surgery, such as gastric bypass that would limit absorption of oral medication.
* Any immunotherapy within 4 weeks of 1st dose of the study.
* Concurrent participation in another therapeutic clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 453 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To establish if combining acalabrutinib with R-CHOP improves efficacy, compared to RCHOP alone, for the treatment of previously untreated patients with DLBCL to a degree that justifies further development of this approach. | Last patient's last follow up, approximately 4.5 years. Patients who do not experience a PFS event will be censored at the date of last follow up.
  Progression-free survival (PFS) is defined as time from registration to progression/death from any cause.

SECONDARY OUTCOMES:
To compare PFS between molecular groups. | Last patient's last follow-up, approximately 4.5 years.
  PFS interaction with cell of origin phenotype (ABC, GCB and unclassifiable).
To compare PFS between treatment groups. | Last patient's last follow-up, approximately 4.5 years.
  PFS interaction with clinical variables, including for example IPI, bulk, components of IPI, age and others to be determined in the SAP.
To compare overall survival (OS) between both treatment and molecular groups. | Last patient's last follow-up, approximately 4.5 years. Patients who do not experience an OS event will be censored at the date of last follow-up.
  Overall survival (OS), defined as time from registration to death from any cause.
To compare event free survival (EFS) between both treatment and molecular groups. | Last patient's last follow-up, approximately 4.5 years. Patients who do not experience an EFS event will be censored at the date of last follow-up.
  Event-free survival (EFS), or time to treatment failure, defined as time from registration to any treatment failure including disease progression, or discontinuation of treatment for any reason.
To compare disease free survival (DFS) between both treatment and molecular groups. | Last patient's last follow-up, approximately 4.5 years. Patients who do not experience a DFS event will be censored at the date of last follow-up.
  Disease-free survival (DFS), defined as time of documentation of disease-free state to disease recurrence or death as a result of lymphoma or acute toxicity of treatment.
To compare time to progression (TTP) between both treatment and molecular groups. | Last patient's last follow-up, approximately 4.5 years. Patients who do not experience a TTP event will be censored at the date of last follow-up.
  Time to progression (TTP), defined as time from registration until documented lymphoma progression or death as a result of lymphoma. Deaths from other causes are censored at the time of death.
To compare duration of response (DoR) between both treatment and molecular groups. | Last patient's last follow-up, approximately 4.5 years. Patients who do not experience a RD event will be censored at the date of last follow-up.
  Response duration (DoR), defined as the time from documentation of response until the documentation of relapse or progression.
To compare overall response rate (ORR) and complete response rate (CR) between both treatment groups. | Complete and overall response rates, as recorded at the end of treatment (up to 21 weeks) .
  Assessment using the Lugano Response Criteria for Malignant Lymphoma.
To assess differences in toxicity between assigned treatments. | At all visits up to 24 months follow-up.
  Evaluation of toxicity according to CTCAE version 5.
To assess differences in quality of life between treatment arms. | At baseline, cycle 2 day 1, cycle 3 day 1, cycle 5 day 1, end of treatment and at 3, 6, 12, 20 and 24 month follow-ups. Each cycle is 21 days.
  Application of the EORTC QLQ-C30 and FACT-Lym questionnaires.

OTHER OUTCOMES:
To explore correlation of molecular characteristics in tumour material to clinical outcomes. | At baseline, cycle 2 day 1, cycle 3 day 1, end of treatment and at 3, 6, 9 and 12 month follow-ups. Each cycle is 21 days.
  Applying the following techniques to FFPE tumour material: mutational panel, FISH analysis, immunohistochemical analysis for dual protein expression of Myc and Bcl2 and dynamic changes in ctDNA and methylation based ctDNA during treatment and follow up.
To explore correlation of baseline PET features including tumour burden and bone marrow involvement to clinical outcomes. | Baseline and end of treatment (up to 21 weeks).
  Tumour burden defined by metabolic tumour volume (MTV) and tumour lesion glycolysis (TLG). Bone marrow involvement defined by focal uptake in the bone marrow higher than liver uptake; diffuse bone marrow uptake higher than liver uptake will be recorded and correlated with bone marrow biopsy results where available (number and location of extranodal sites).
To explore combination(s) of clinical risk factors, molecular characteristics and PET features to clinical outcomes. | Baseline and end of treatment (up to 21 weeks).
To compare metabolic response between molecular groups. | Baseline and end of treatment (up to 21 weeks).
To update existing metabolic response criteria using advanced PET reconstructions. | Baseline and end of treatment (up to 21 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, Principal Investigator — University of Southampton
Locations (33):
- United Kingdom (33):
  - Colchester General Hospital, Colchester, Essex
  - East Kent Hospitals NHS Foundation Trust, Canterbury, Kent
  - Monklands Hospital, Airdrie
  - Victoria Hospital, Blackpool
  - University Hospital Dorset NHS Foundation Trust (Bournemouth and Poole Hospitals), Bournemouth
  - Queens Hospital, Burton-on-Trent
  - Addenbrooke's Hospital, Cambridge
  - Royal Derby Hospital, Derby
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Ipswich Hospital, Ipswich
  - St James Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Chase Farm and Barnet Hospitals, London
  - Lewisham and Greenwich NHS Trust, London
  - University College London Hospital, London
  - Maidstone Hospital, Maidstone
  - The Christie Hospital, Manchester
  - Milton Keynes University Hospital, Milton Keynes
  - Freeman Hospital, Newcastle
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Royal Oldham Hospital, Oldham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Queen's Hospital, Romford
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Singleton Hospital, Swansea
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Worthing and St Richards Hospitals, Worthing

IPD SHARING:
Plan to Share IPD: No